CLINICAL TRIAL: NCT00936377
Title: A Randomized, Double-Blind, Placebo Controlled, Dose Escalation Study of Dexmedetomidine as Adjunctive Therapy for Alcohol Withdrawal
Brief Title: Dexmedetomidine as Adjunctive Therapy for Alcohol Withdrawal
Acronym: DATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-0406
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Acute Alcohol Withdrawal
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexmedetomidine, low dose (Experimental): Dexmedetomidine 0.4 µg/kg per hour administered for a maximum duration of five days
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine, high dose (Experimental): Dexmedetomidine 1.2 µg/kg per hour administered for a maximum duration of five days
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine at 0.4 or 1.2 µg/kg per hour is administered for a maximum duration of five days
  Other Names: Precedex
  Arms: Dexmedetomidine, high dose; Dexmedetomidine, low dose
Other: Placebo — Normal saline for five days.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate dexmedetomidine as adjunctive therapy of severe alcohol withdrawal of medical ICU patients. Specifically, this study will assess whether adjunctive dexmedetomidine reduces the doses of conventional agents used for alcohol withdrawal while maintaining patient comfort and safety and will explore if dexmedetomidine exhibits a dose-dependent profile of action when it is used for this indication. In addition, this study will assess the relationships between alcohol withdrawal, therapy with dexmedetomidine, and potential serum biomarkers of alcohol withdrawal.

DETAILED DESCRIPTION:
The objectives of this randomized, double-blind, placebo controlled, dose escalation study are a) to determine if adding dexmedetomidine to symptom-triggered, standard therapy of severe alcohol withdrawal reduces the dose requirements of conventional sedatives, analgesics, and neuroleptics; maintains patient comfort and safety; and prevents and shortens tracheal intubation; b) to explore whether dexmedetomidine acts in a dose-dependent manner to reduce the dose requirements of conventional sedatives, analgesics, and neuroleptics while maintaining patient comfort; and c) determine the association between alcohol withdrawal and potential serum biomarkers of alcohol withdrawal and assess whether these are expressed differently when dexmedetomidine is used as adjunctive therapy. Dexmedetomidine will be added to existing sedative therapies in an effort to decrease the use of these agents while maintaining patient comfort. The study will randomize twenty-four patients in a double-blind manner to receive placebo or dexmedetomidine at doses of 0.4 or 1.2 µg/kg per hour for a maximum duration of five days. All patients will be managed using an existing institution-specific, symptom-triggered alcohol withdrawal protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Severe alcohol withdrawal defined by a CIWA score ≥ 15 and the need for at least 16 mg of lorazepam over a four-hour period. All lorazepam doses, whether oral or intravenous, will contribute to the cumulative amount.
2. Patients receiving standard therapy for severe alcohol withdrawal according to a symptom-triggered alcohol withdrawal protocol. Lorazepam is the preferred benzodiazepine agent for patients requiring ICU admission due to alcohol withdrawal.
3. Informed consent within 36 hours of qualifying for the study.

Exclusion Criteria:

1. Patients < 18 years of age or > 85 years of age.
2. Patients receiving benzodiazepine therapy for purposes other than alcohol withdrawal (e.g. sedation).
3. Patients with alcohol withdrawal not requiring ICU admission.
4. Patients receiving epidural administration of medication(s).
5. Comatose patients by metabolic or neurologic affectation.
6. Patients with active myocardial ischemia or second- or third-degree heart block.
7. Moribund state with planned withdrawal of life support.
8. Patients with known or suspected severe adverse reactions to dexmedetomidine (or clonidine).
9. Pregnant females or females suspected of being pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert MacLaren, PharmD, Principal Investigator — University of Colorado School of Pharmacy
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Derived] Reynolds PM, Mueller SW, MacLaren R. A comparison of dexmedetomidine and placebo on the plasma concentrations of NGF, BDNF, GDNF, and epinephrine during severe alcohol withdrawal. Alcohol. 2015 Feb;49(1):15-9. doi: 10.1016/j.alcohol.2014.11.006. Epub 2015 Jan 22. PMID 25638740
- [Derived] Mueller SW, Preslaski CR, Kiser TH, Fish DN, Lavelle JC, Malkoski SP, MacLaren R. A randomized, double-blind, placebo-controlled dose range study of dexmedetomidine as adjunctive therapy for alcohol withdrawal. Crit Care Med. 2014 May;42(5):1131-9. doi: 10.1097/CCM.0000000000000141. PMID 24351375

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Full Range); unit: years] | 47 [28 to 60] | 50 [30 to 56] | 51 [30 to 61] | 49.3 [28 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 8 | 7 | 7 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 5 | 7 | 4 | 16
  Other | 3 | 1 | 4 | 8
Weight [Mean (Full Range); unit: kg] | 87.1 [44.5 to 126] | 84.5 [60 to 126] | 81.5 [58 to 98] | 84.4 [44.5 to 126]
Acute Physiologic And Chronic Health Evaluation (APACHE) III [Mean (Inter-Quartile Range); unit: units on a scale] — APACHE III measures the severity of disease for adult patients admitted to intensive care units. The point score is calculated as a summation from scores assigned to a patient's age, primary comorbidity, preexisting comorbidities, location prior to ICU admission, Glasgow Coma Scale, and 20 routine physiological measurements. APACHE III scores range from 0 to 299. This provides an initial risk classification of severely ill hospitalized patients in defined groups with higher scores indicating greater disease severity and correlated to higher mortality risk.
  units on a scale | 69.5 [65 to 72] | 56.5 [43 to 64] | 49.5 [30 to 68] | 58.5 [30 to 72]
Endotracheal Intubation at Study Entry [Number; unit: participants]
  Intubated | 5 | 3 | 5 | 13
  Not intubated | 3 | 5 | 3 | 11
Child-Pugh Score [Mean (Full Range); unit: units on a scale] — The Child-Pugh score is used to assess the prognosis of chronic liver disease. The point score is calculated from the summation of points assigned for total bilirubin (serum), albumin (serum), prothrombin time, and the presence of ascites and encephalopathy. The range is from 0 to 15. Grade A liver disease (scores of 5-6) predict two-year survival of 85%. Grade B liver disease (scores of 7-9) predict two-year survival of 55%. Grade C liver disease (scores of 10-15) predict two-year survival of 35%.
  units on a scale | 7 [6 to 9] | 6 [6 to 9] | 6 [5 to 11] | 6.3 [5 to 11]
Lorazepam requirement 24 Hour Prior to Study Entry [Mean (Inter-Quartile Range); unit: mg] | 94 [52 to 148] | 75 [28 to 190] | 39 [31 to 91] | 69.3 [28 to 190]
Time from Study Qualification to Study Drug Start [Median (Inter-Quartile Range); unit: hours] | 17.1 [6.5 to 33.7] | 13.5 [3.4 to 27] | 10.4 [1.7 to 19.9] | 14 [1.7 to 33.7]

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Lorazepam Dose Over the First Seven Days of Alcohol Withdrawal
Time Frame: Seven days
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8
mg | 180.5 [79.3 to 223.4] | 112.5 [48.8 to 746.8] | 109.1 [40.9 to 227.4]
Statistical Analysis 1: Comparison: Dexmedetomidine, Low Dose vs Placebo; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexmedetomidine, High Dose vs Placebo; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in 12-Hour Lorazepam Requirement Pre- and Post-Treatment
Time Frame: 12 hours before treatment, 12 hours after treatment on first day of starting study drug
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8
mg | -42.5 [-52.7 to -1.6] | -34.3 [-61.9 to -14.5] | -17.5 [-24.3 to 36.7]
Statistical Analysis 1: Comparison: Dexmedetomidine, Low Dose vs Placebo; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexmedetomidine, High Dose vs Placebo; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in 24-Hour Lorazepam Requirement Pre- and Post-Treatment
Time Frame: 24 hours before treatment, 24 hours after treatment on first day of starting study drug
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8
mg | -62.1 [-118 to -8.8] | -45 [-68.9 to -16.8] | -8 [-31.3 to 76.2]
Statistical Analysis 1: Comparison: Dexmedetomidine, Low Dose vs Placebo; Test type: Superiority or Other; p = 0.066, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexmedetomidine, High Dose vs Placebo; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: The Degree of Alcohol Withdrawal Assessed by Clinical Institute Withdrawal Assessment (CIWA) Scores
Description: Proportion of clinical institute withdrawal assessment (CIWA) Scores listed as severe or moderate 24 Hours after Starting Study Drug. All subjects had at least four CIWA assessments.The CIWA is a ten item scale with each item on the scale scored independently on a 0-7 or 0-4 scale, and the summation of the scores yielding an aggregate value that correlates to the severity of alcohol withdrawal. Ranges of scores are from 0 to 67. Mild alcohol withdrawal is defined with a score less than or equal to 15, moderate with scores of 16 to 20, and severe with any score greater than 20. The ten items evaluated include nausea and vomiting, tremor, sweats, anxiety, agitation, tactile disturbances, auditory disturbances, visual disturbances, headache, and orientation.
Time Frame: Every 2-4 hours for 24 hours after starting study drug
Measure: Number; unit: percentage of ciwa assessment
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8
percentage of ciwa assessment
  severe | 11 | 15 | 25
  moderate | 31 | 24 | 22
Statistical Analysis 1: Comparison: Dexmedetomidine, Low Dose vs Placebo; Percentage of CIWA scores rates as severe; Test type: Superiority or Other; p = 0.18, Chi-squared, Corrected — Percentage of CIWA scores rates as severe
Statistical Analysis 2: Comparison: Dexmedetomidine, High Dose vs Placebo; Test type: Superiority or Other; p = 0.35, Chi-squared, Corrected — Percentage of CIWA scores rates as severe

5. Secondary Outcome: The Occurrence of Adverse Events.
Description: Occurrence of hypotension or bradycardia while on study drug
Time Frame: Seven days
Measure: Number; unit: participants
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8
participants
  Hypotension | 1 | 2 | 0
  Bradycardia | 1 | 3 | 0
Statistical Analysis 1: Comparison: Dexmedetomidine, Low Dose vs Placebo; For hypotension; Test type: Superiority or Other; p = 1, Fisher Exact
Statistical Analysis 2: Comparison: Dexmedetomidine, High Dose vs Placebo; For hypotension; Test type: Superiority or Other; p = 0.47, Fisher Exact
Statistical Analysis 3: Comparison: Dexmedetomidine, Low Dose vs Placebo; For bradycardia; Test type: Superiority or Other; p = 1, Fisher Exact
Statistical Analysis 4: Comparison: Dexmedetomidine, High Dose vs Placebo; For bradycardia; Test type: Superiority or Other; p = 0.2, Fisher Exact

6. Secondary Outcome: Plasma Epinephrine Concentrations Across Groups Over Time
Description: Plasma epinephrine concentrations
Time Frame: Four days with samples measured prior to study drug and 48 and 96 hours after starting study drug
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8
ng/mL
  Baseline | 0.27 (0.17) | 0.29 (0.1) | 0.31 (0.25)
  Time 48 hours | 0.27 (0.47) | 0.21 (0.09) | 0.27 (0.17)
  Time 96 hours | 0.26 (0.33) | 0.27 (0.17) | 0.3 (0.04)
Statistical Analysis 1: Comparison: Dexmedetomidine, High Dose; Test type: Superiority or Other; p < 0.05, Repeated measures ANOVA

7. Secondary Outcome: Duration of Study Drug Administration
Time Frame: The duration of study drug in hours as measured when the subject was discharged from the ICU, for up to 24 weeks
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8
hours | 53.1 [39.4 to 89.5] | 78 [22.1 to 112.5] | 70.3 [25 to 120]
Statistical Analysis 1: Comparison: Dexmedetomidine, Low Dose vs Placebo; Test type: Superiority or Other; p = 0.5, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexmedetomidine, High Dose vs Placebo; Test type: Superiority or Other; p = 0.95, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: ICU Length of Stay
Time Frame: The duration of ICU stay in days as measured at time of hospital discharge, for up to 24 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8
days | 5.5 [2.5 to 9.9] | 3.8 [2.4 to 10] | 4 [1.9 to 7.1]
Statistical Analysis 1: Comparison: Dexmedetomidine, Low Dose vs Placebo; Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexmedetomidine, High Dose vs Placebo; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine, Low Dose | Dexmedetomidine, High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine, Low Dose (N=8) | Dexmedetomidine, High Dose (N=8) | Placebo (N=8)
Hypotension (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Hypertension (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No